CLINICAL TRIAL: NCT04867473
Title: Teleyoga for Lyme Disease
Brief Title: Feasibility of Teleyoga for Treatment of Lyme Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Peter Bayley, Investigator, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 49667
Record Dates: First submitted 2021-04-16; First posted 2021-04-30 (Actual); Results first posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2023-08

CONDITIONS: Lyme Disease
Keywords: yoga; telehealth; chronic pain
MeSH Terms: conditions — Lyme Disease; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Participants will attend teleyoga sessions once per week, with assessments at beginning and end of treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Teleyoga (Experimental): Lyme disease participants will attend home-based yoga sessions using HIPAA-compliant telehealth software and devices and complete pain inventory questionnaires pre and post-treatment
  Interventions: Behavioral: Teleyoga

INTERVENTIONS:
Behavioral: Teleyoga — 12 weekly 75 minute therapist-led teleyoga sessions

SUMMARY:
Primary Aims: Modify an existing teleyoga intervention to use with Lyme disease (LD) patients and address the technical challenges of at-home teleyoga

DETAILED DESCRIPTION:
Participants with symptoms of Lyme disease (n=15) will participate individually in a weekly tele-yoga class using an iPad loaned by the study. Participants will choose where to attend these remote treatment sessions. Yoga treatment will last 12 weeks. Participants' subjective pain will be rated at baseline and end-of-treatment using a standard pain scale. Also assessed will be participant adherence to study protocol by tracking treatment attendance

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable Lyme disease
* Has not begun new pain medications or other treatments in the last month
* English literacy
* Wireless internet connection at home

Exclusion Criteria:

* Participation in another concurrent clinical trial
* Back surgery within the last 12 months
* Unstable, coexisting mental illness or psychiatric condition
* Active, current suicidal intent or plan
* Attended or practiced yoga ≥ 1 x in the past 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2022-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Bayley, Ph.D., Study Director — VA Palo Alto Health Care System and Stanford University; Jerome A Yesavage, M.D., Principal Investigator — Stanford University and VA Palo Alto Health Care System
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 1:1 Sessions: Yoga will be delivered in either a 1-on-1 format between the yoga therapist and the participant.
  Participants will receive at-home teleyoga classes via video conferencing.
- Group Sessions: Yoga will be delivered in a group format between the yoga therapist and the participant.
  Participants will receive at-home teleyoga classes via video conferencing.
Period: Overall Study
Arm/Group | 1:1 Sessions | Group Sessions
Started | 5 | 10
Completed | 5 | 8
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1:1 Sessions | Group Sessions | Total
Number analyzed (Participants) | 5 | 10 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 2 participants dropped out in the group format
  years
    number analyzed (Participants) | 5 | 8 | 13
    (all) | 39 (14.3) | 43.5 (12.6) | 41.3 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 2 participants dropped out in the group format
  Participants
    number analyzed (Participants) | 5 | 8 | 13
    Female | 4 | 8 | 12
    Male | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 2 participants dropped out in the group format
  Participants
    number analyzed (Participants) | 5 | 8 | 13
    American Indian or Alaska Native | 0 | 2 | 2
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 5 | 6 | 11
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — Population: 2 participants dropped out in the group format
  Participants
    United States: number analyzed (Participants) | 5 | 8 | 13
    United States | 5 | 8 | 13

OUTCOME MEASURES:

1. Primary Outcome: Change of Pain Score From Baseline
Description: Scores on the Pain, Enjoyment, General Activity (PEG) Scale; with values from 0 to 10 and higher scores indicating worse outcomes
Time Frame: Measured at baseline and again at the end of 12 weeks of treatment
Population: 2 dyads dropped out
Measure: Number; unit: score on a scale
Arm/Group | 1:1 Sessions | Group Sessions
Number analyzed (Participants) | 5 | 8
score on a scale
  Average PEG Score at Baseline | 5.7 | 4.8
  Average PEG score at end of treatment | 2.9 | 4.6

2. Secondary Outcome: Adherence to the Treatment Protocol
Description: Percentage of participants who attend ≥65 percent of treatment sessions; values range from 0 percent to 100 percent with higher percentages indicative of a better outcome
Time Frame: at study completion, an average of 7 months
Measure: Count of Participants; unit: Participants
Arm/Group | 1:1 Sessions | Group Sessions
Number analyzed (Participants) | 5 | 8
Participants | 5 | 7

ADVERSE EVENTS:
Time Frame: baseline to end of treatment (12 weeks)
Arm/Group | 1:1 Sessions | Group Sessions
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/10
Other Adverse Events (participants affected / at risk) | 0/5 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-06-21): https://cdn.clinicaltrials.gov/large-docs/73/NCT04867473/Prot_SAP_ICF_000.pdf